CLINICAL TRIAL: NCT02200042
Title: Randomized Phase III Study of Focal Radiation Therapy for Unresectable, Localized Intrahepatic Cholangiocarcinoma
Brief Title: Radiation Therapy vs. Observation Following Gemcitabine and Cisplatin for Inoperable Localized Liver Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI001; NCI-2014-00849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PNRG-GI001_A02PAMDREVW01; PNRG-GI001_A01PAMDREVW01; NRG-GI001 (Other: NRG Oncology); NRG-GI001 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-07-08; First posted 2014-07-25 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Stage III Intrahepatic Cholangiocarcinoma; Stage IVA Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Intervention Model Description: Randomization ratio (Experimental:Observation) = 2:1
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation therapy (Experimental): Liver-directed radiation therapy
  Interventions: Radiation: Image Guided Radiation Therapy
- Observation (No Intervention): No radiation therapy

INTERVENTIONS:
Radiation: Image Guided Radiation Therapy — Patients undergo 15 fractions of image-guided radiation therapy delivered over 19-26 or 27-34 days.
  Other Names: IGRT; image-guided radiation therapy
  Arms: Radiation therapy

SUMMARY:
This randomized phase III trial studies how well gemcitabine hydrochloride and cisplatin with or without radiation therapy work in treating patients with localized liver cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x rays to kill tumor cells. It is not yet known whether giving gemcitabine and cisplatin is more effective with or without radiation therapy in this patient population. Patients register to this study after receiving gemcitabine and cisplatin.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the addition of liver-directed radiation therapy with respect to overall survival (OS) for patients with unresectable, localized intrahepatic cholangiocarcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the addition of liver-directed radiation therapy with respect to local control for patients with unresectable, localized intrahepatic cholangiocarcinoma.

II. To evaluate the addition of liver-directed radiation therapy with respect to adverse events for patients with unresectable, localized intrahepatic cholangiocarcinoma.

III. To evaluate the addition of liver-directed radiation therapy with respect to regional control for patients with unresectable, localized intrahepatic cholangiocarcinoma.

IV. To evaluate the addition of liver-directed radiation therapy with respect to distant metastases for patients with unresectable, localized intrahepatic cholangiocarcinoma.

V. To evaluate the addition of liver-directed radiation therapy with respect to progression-free survival for patients with unresectable, localized intrahepatic cholangiocarcinoma.

After completion of study treatment, patients are followed up every 3 months for 3 years then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of intrahepatic cholangiocarcinoma (IHC) without distant extrahepatic metastasis prior to study entry. Patients with an adenocarcinoma suggestive of a pancreaticobiliary primary with radiographic findings consistent with an intrahepatic cholangio-carcinoma are eligible.
2. Patient must have 1 lesion with a maximum AXIAL diameter of 12cm at the time of study entry. Up to 3 satellite lesions are permitted. Satellite lesions, are defined as lesions less than 2 cm that are within 1 cm of the periphery of the dominant lesion (gross tumor volume [GTV]) are permitted. The satellite lesions are NOT included in the AXIAL diameter measurement. Regional Lymph Node involvement within the porta hepatis (as medial as superior mesenteric vein [SMV] portal vein confluence) is permitted if nodes are deemed clinically positive (i.e. FDG [Fluorine 18 fluorodeoxyglucose] avid);
3. Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

   • Pre-study entry Scan (REQUIRED for All Patients to confirm no progression): computed tomography (CT) scan chest/abdomen/pelvis with multiphasic liver CT scan within 30 days prior to study entry. If CT contrast is contraindicated, CT chest without contrast and MRI of abdomen and pelvis is permitted;
4. Zubrod Performance Status 0-1 at the time of study entry;
5. Age ≥ 18;
6. Complete blood count (CBC) / differential obtained within 21 days prior to study entry, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3;
   * Platelets ≥ 75,000 cells/mm3;
   * Total bilirubin < 2.5 mg/dl;
   * Aspartate Aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (Serum glutamic pyruvic transaminase [SGPT]) < 5.0 X institutional upper limit of normal;
   * Albumin ≥ 2.5mg/dl;
   * Creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for subject with creatinine levels above institutional normal;
   * Hemoglobin(Hgb) ≥ 9.0 g/dl. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable.)
7. Patient must provide study specific informed consent prior to study entry;
8. Negative Beta-Human Chorionic Gonadotropin (bHCG) prior to study entry if patient is pre or peri-menopausal.
9. Must have received 6 months of Gemcitabine/Cisplatin chemotherapy without progression. Disease response to chemotherapy is also permitted. If toxicity precludes 6 months of chemotherapy at least 4 months of Gemcitabine/Cisplatin must have been administered.

Exclusion Criteria:

1. Multiple lesions that don't meet the criteria as satellite lesions as defined in protocol;
2. Extrahepatic metastases or malignant nodes beyond the periportal region. Celiac, pancreaticoduodenal and para-aortic nodes> 2 cm are ineligible. Note that benign non-enhancing periportal lymphadenopathy is not unusual in the presence of hepatitis and is permitted, even if the sum of enlarged nodes is > 2.0 cm;
3. Hepatic insufficiency resulting in clinical jaundice, encephalopathy and/or variceal bleed at the time of study entry;
4. Prior radiotherapy to the region of the liver that would result in overlap of radiation therapy fields;
5. Prior selective internal radiotherapy/hepatic arterial Yttrium therapy, at any time;
6. Direct tumor extension into the stomach, duodenum, small bowel or large bowel;
7. Prior invasive malignancy, excluding the current diagnosis, (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years. (Note: carcinoma in situ of the breast, oral cavity, or cervix is all permissible);
8. Prior systemic chemotherapy for the study cancer other than gemcitabine/cisplatin; note that prior chemotherapy for a different cancer is allowable;
9. Currently receiving other anti-cancer agents;
10. Participants who require anticoagulation should receive low-molecular weight or standard heparin and not warfarin;
11. Prior surgery for the IHC. (Liver resection is not allowed);
12. Severe, active co-morbidity, defined as follows:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months of study entry;
    * Transmural myocardial infarction within the last 6 months of study entry;
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study entry;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to study entry;
    * HIV positive with CD4 (cluster of differentiation 4) count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter at the time of study entry. Note also that HIV testing is not required for eligibility for this protocol;
    * End-stage renal disease (ie, on dialysis or dialysis has been recommended).
13. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic;
14. Grade 3 or higher peripheral neuropathy at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Hong, Principal Investigator — NRG Oncology
Locations (34):
- United States (33):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Medical Center Sacramento, Sacramento, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - ProCure Proton Therapy Center-Seattle, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Tao R, Krishnan S, Bhosale PR, Javle MM, Aloia TA, Shroff RT, Kaseb AO, Bishop AJ, Swanick CW, Koay EJ, Thames HD, Hong TS, Das P, Crane CH. Ablative Radiotherapy Doses Lead to a Substantial Prolongation of Survival in Patients With Inoperable Intrahepatic Cholangiocarcinoma: A Retrospective Dose Response Analysis. J Clin Oncol. 2016 Jan 20;34(3):219-26. doi: 10.1200/JCO.2015.61.3778. Epub 2015 Oct 26. PMID 26503201

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy: Liver-directed radiation therapy
  Radiation Therapy: Patients undergo 15 fractions of image-guided radiation therapy delivered over 19-26 or 27-34 days.
Period: Overall Study
Arm/Group | Radiation Therapy | Observation
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients with baseline data
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy | Observation | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival time is defined as time from randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been on study for at least two years.
Population: No patients have outcome data.
Arm/Group | Radiation Therapy | Observation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Distant Metastases
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been on study for at least two years.
Population: No patients have outcome data.
Arm/Group | Radiation Therapy | Observation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Adverse Events Evaluated Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been on study for at least two years.
Population: No patients have outcome data.
Arm/Group | Radiation Therapy | Observation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Local Progression
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been on study for at least two years.
Population: No patients have outcome data.
Arm/Group | Radiation Therapy | Observation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been on study for at least two years.
Population: No patients have outcome data.
Arm/Group | Radiation Therapy | Observation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Regional Progression Defined as Progression or Existing or Appearance of New Nodal Disease
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been on study for at least two years.
Population: No patients have outcome data.
Arm/Group | Radiation Therapy | Observation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No adverse event data was collected on this study due to early termination.
Description: No adverse event data was collected on this study due to early termination.
Arm/Group | Radiation Therapy | Observation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 1 subject accrued out of 146 planned. The registered subject withdrew consent the same day as randomization and therefore has no outcome data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02200042/Prot_SAP_000.pdf